CLINICAL TRIAL: NCT02060747
Title: Optimization of Osteoporosis Management Among Patients Older Than 45 Years Old With Low Energy Fracture.
Acronym: OPTIPOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OPTIPOST
Record Dates: First submitted 2014-01-27; First posted 2014-02-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-12

CONDITIONS: Osteoporosis, Management Care, Fracture
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coordinator-based post fracture program (Experimental): The intervention arm deals with the intervention of a nurse trained in the management of osteoporosis fractures assisted by a clinical research technician who will manage the logistics and reglementary aspects of the study (patient enrollment, quality and study proceedings).
  Interventions: Behavioral: Coordinator-based post fracture program
- standard care (No Intervention)

INTERVENTIONS:
Behavioral: Coordinator-based post fracture program
  Arms: Coordinator-based post fracture program

SUMMARY:
Harrington's metaphorical depiction captures the essence of the problem : "Osteoporosis care of fracture patients has been characterized as the Bermuda Triangle made up of orthopaedists, primary care physicians and osteoporosis experts into which the fracture patient disappears".

The most effective way to achieve this goal is through implementation of coordinator-based post fracture models of care. Exemplar models have been refered to as "Fracture Liaison Service" (United-Kingdom [1-3], Europe [4,5] and Australia [6-8]) "Osteoporosis Coordinator Program" (Canada [9,10]) or "Care Manager Programs" (USA [11,12]).

The objective of this trial is to assess efficacy of a new coordinator-based post-fracture program in the Saint-Joseph Hospital in Paris to improve the management of osteoporosis after fracture thanks to an optimal recommendations practice to reduce the incidence of secondary fractures.

Men and women are included aged over 45 years with fragility wrist and hip fractures.

Evaluation criteria are based on the evidence-based assessment (stratify risk, identify secondary causes of osteoporosis, fracture evaluation), the medication adherence, others prescriptions adherence (osteodensitometry), the incidence of secondary fractures and number of falls.

Number of patients : 200 Duration of the study: 3 years Patients' participation duration: 6 months

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 45 years
* Fragility wrist and hip fractures
* Volunteer

Exclusion Criteria:

* Public route accident
* Emergency illness associated
* Short life expectancy
* Not volunteer
* Bedridden patient

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patient with a correct management care. | 6 months
  This outcome is a composite outcome wich differ with each fracture type. It will be assess 6 months after patient inclusion.
  An adequate management care is defined for each fracture as below.
  * For wrist fracture: medical visit at J15, osteodensitometry, therapeutic decision if necessary (if not, reasons have to be precised in medical sheet).
  * For hip fracture: osteodensitometry if necessary, therapeutic (chronic care) decision if necessary (if not, reasons have to be precised in medical sheet).

SECONDARY OUTCOMES:
Patient adherence to their osteoporosis medication (Morisky composite score) and exploration (osteodensitometry). | 6 months

OTHER OUTCOMES:
Number of rehospitalisation for fracture. | 6 months
Number of falls over 6 months post-inclusion. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Mc Lellan AR and al. Osteoprosis Int. 2003; 1028-1034 2. Wright SA and al. Rheumatol Int 2005; 489-490 3. Clunie G and al. J Orthop Nurs 2008; 156-162 4. Boudou L and al. Osteoporos Int 2011; 2099-2016 5. Huntjzens KM ana al. Osteoporos Int 2011; 2119-2135 6. Cooper MS and al. Osteoporos Int 2012; 97-107 7. Inderjeeth CA and al. Med J Aus 2010; 149-153 8. Lih A and al. Osteoporos Int 2011; 849-858 9. Bogoch ER and al. J Bone Joint Surg Am 2006; 25-34 10. SAbder B abd al. J Bone Joint Surg Am 2008; 1197-1205 11. Dell R and al. J Bone Joint Surg Am 2008; 188-194 12. Greene D and al. J Am Acad Nurse Pract 2010; 326-329